CLINICAL TRIAL: NCT02031380
Title: Improving Ophthalmic Medication Adherence
Brief Title: iDropper Usability in Glaucoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Care Team Solutions (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R43EY023122-01A1-1; 1R43EY023122-01A1 (NIH)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Glaucoma, Open-Angle [C11.525.381.407]
Keywords: Glaucoma; Open angle glaucoma; ocular hypertension; compliance
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open angle glaucoma - iDropper device (Experimental): Device
  Interventions: Device: Open angle glaucoma - iDropper device

INTERVENTIONS:
Device: Open angle glaucoma - iDropper device — The iDropper system is an eye drop dispensing device and medication monitor designed to optimize adherence behaviors for glaucoma patients.

SUMMARY:
The purpose of this study is to evaluate the usability of a medication management support system for glaucoma patients self-administering eye drops named iDropper. The iDropper system is a home-based ocular medication management system that reminds, instructs, dispenses, and records eye drop medication usage. The iDropper system will be evaluated among a cohort of glaucoma subjects self-administering eye drops for 4-weeks.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of vision loss in the United States, impacting the lives of ~4 million people. Left untreated or inadequately managed, it causes blindness -- the second ranking cause of blindness in the world as well as the leader among African Americans. Estimates project 79.6 million glaucoma diagnoses worldwide by 2020; of these, 74% will have open-angle glaucoma (OAG), which occurs virtually without symptoms. The explanation for such strikingly high disease prevalence and blindness rates is partially due to the asymptomatic nature of glaucoma. However, deficient adherence to glaucoma ocular hypotensive drops is a significant and escalating health care problem.

Glaucoma eye drops are often the first therapeutic choice and very effective at controlling intraocular pressure (IOP) to prevent eye damage. However, glaucoma is a chronic condition and daily dosing regimens for medications can be complex and difficult to manage with impaired vision. Consequently, adherence and persistence to glaucoma eye drop regimens over time becomes quite poor. Overwhelming research brings the unwelcome conclusion that long term persistence with glaucoma medication is 33-39% at one year and positively contributes to blindness.

Currently, no mechanism exists for supporting and monitoring glaucoma eye drop compliance.

The purpose of this study is to evaluate the usability of a medication management support system for glaucoma patients self-administering eye drops named iDropper. The iDropper system is a home-based ocular medication management system that reminds, instructs, dispenses, and records eye drop medication usage. The iDropper system will be evaluated among a cohort of glaucoma subjects self-administering eye drops for 4-weeks.

At study conclusion usability and satisfaction assessments will be performed to evaluate iDropper system performance.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age;
* Physician diagnosis of: open angle glaucoma, angle-closure glaucoma, glaucoma suspect, or ocular hypertension
* Responsible for self-administration of eye drops.
* No surgery within the prior 3 months;
* Able to speak and read English;

Exclusion Criteria:

* Having any concurrent medical or psychiatric condition that, in the investigator's opinion, may preclude participation in this study; or
* Cognitive or visual impairment that would interfere with completing a self-administered questionnaire.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Usability questionnaire | 4 weeks after trial start
  Written questionnaire assessing usability of the iDropper system by participants

SECONDARY OUTCOMES:
Satisfaction questionnaire | 4 weeks after study start
  Questionnaire assessing participant satisfaction with features of the iDropper system.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bailey, PhD, Study Director — Care Team Solutions; Steven Chalfin, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Background] Congdon N, O'Colmain B, Klaver CC, Klein R, Munoz B, Friedman DS, Kempen J, Taylor HR, Mitchell P; Eye Diseases Prevalence Research Group. Causes and prevalence of visual impairment among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):477-85. doi: 10.1001/archopht.122.4.477. PMID 15078664
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940